CLINICAL TRIAL: NCT04920110
Title: Validation of the Observer-Reported Communication Ability (ORCA) Measure in Rett Syndrome
Brief Title: Development of the ORCA Communication Measure for Rett Syndrome
Acronym: Rett-ORCA
Status: Completed | Type: Observational
Sponsor: Rett Syndrome Research Trust (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: ORCA-101-RSRT
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Rett Syndrome
Keywords: ORCA; Communication; Duke; MECP2; RSRT
MeSH Terms: conditions — Rett Syndrome; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: Qualitative Interviews: Approximately 20 parents/caregivers will discuss typical communication abilities of their loved one and complete the ORCA measure for determination of its content validity through a hybrid approach of concept elicitation and cognitive testing.
- Phase 2: Cross-Sectional Assessment of Psychometric Properties: Approximately 250 parents/caregivers will complete the ORCA measure and additional measures to determine its psychometric properties including reliability, floor/ceiling effects and construct validity.

SUMMARY:
This measurement validation study will use qualitative and quantitative methodology to evaluate the Observer-Reported Communication Ability Measure (ORCA), to appropriately capture communication abilities in individuals with Rett syndrome. The ORCA Measure is a caregiver-reported questionnaire that collects caregiver observations of their child's communication abilities including expressive, receptive and pragmatic communication types. Caregivers will participate via phone interviews and online surveys. Approximately 270 participants will be enrolled.

DETAILED DESCRIPTION:
This study will develop the Observer-Reported Communication Ability Measure (ORCA), originally validated for Angelman syndrome, to appropriately capture communication abilities in individuals with Rett syndrome. The ORCA Measure is a caregiver-reported questionnaire that collects caregiver observations of their child's communication abilities including expressive, receptive and pragmatic communication. The goal of the study is to generate a validated tool to comprehensively assess communication in Rett syndrome and create an important endpoint for use in clinical trials.

In phase 1, a hybrid approach to concept elicitation and cognitive testing will occur with caregivers to assess the existing ORCA measure and evaluate ORCA content validity. Approximately 20 parents/caregivers of individuals with Rett syndrome will participate in qualitative in-depth interviews. The ORCA measure, instructions, recall period, and response choices will be evaluated.

In phase 2, psychometric properties including reliability, floor/ceiling effects, construct validity, and test-retest will be evaluated with approximately 250 caregiver-parents of individuals with Rett syndrome. Caregivers will also complete additional questionnaires to allow comparison between the ORCA measure and existing measures. Analysts will use a variety of statistical methods to evaluate the psychometric properties of the ORCA measure in Rett syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Parent or caregiver at least 18 years of age, with a female child, age 2 or older, diagnosed with Rett syndrome confirmed by a disease-causing MECP2 genetic mutation.
* Fluency in the English language
* Currently lives with the child with Rett syndrome
* Ability and willingness to participate in all study activities.
* Access to a telephone and/or access to a device with internet access that is capable of supporting electronic survey completion

Exclusion Criteria:

* Parent or caregiver with clinically significant condition or situation that makes them not be suitable for the study, in the opinion of research staff.
* Parent or caregiver of a child with Rett syndrome who also has another diagnosis in addition to Rett syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents/caregivers of individuals with Rett syndrome confirmed by an MECP2 genetic mutation, who are fluent in English.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Observer-Reported Communication Ability Measure (ORCA) | 1 year
  Using qualitative and quantitative methodology the existing ORCA measure will be evaluated for use in Rett syndrome and modified if needed. The ORCA measure produces a single score that is an estimate of an individual's overall level of communication ability. Higher ORCA scores reflect greater communication ability; the mastery of expressive, receptive, and pragmatic types of communication and higher vocabularies for verbal words and symbols on assistive devices. The ORCA T-score range is from 26.82 to 83.24.

CONTACTS AND LOCATIONS:
Overall Officials: Bryce B Reeve, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No